CLINICAL TRIAL: NCT02830893
Title: Lever Actuated Rehabilitation of the Arm Using Wheelchair Propulsion and Computer Gaming
Brief Title: Efficacy Study of the LARA Wheelchair System for Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, Professor of Neurology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-3304
Record Dates: First submitted 2016-07-05; First posted 2016-07-13 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- The LARA Therapy (Experimental): The LARA arm of this study will use the LARA system while study participants are staying at the acute rehabilitation unit of UC Irvine Douglas Hospital. LARA is a system that facilitates patients to perform high amounts of arm movement with the affected upper extremity. Study participants are able to actively propel themselves in the unit.
  Interventions: Device: LARA
- The Standard Therapy (Active Comparator): The control arm of this study will use a standard wheelchair while study participants are staying at the acute rehabilitation unit of UC Irvine Douglas Hospital. Study participants will have no exposure to LARA and they will use a standard wheelchair. They will use their unaffected upper and lower extremities to propel themselves in the unit.
  Interventions: Behavioral: Standard

INTERVENTIONS:
Device: LARA — Study participants will use LARA to propel themselves and to play computer games with the impaired upper extremity for 30 min/day in addition to standard of care rehabilitation therapy for 3 weeks or the duration of their stay.
  Arms: The LARA Therapy
Behavioral: Standard — Study participants will receive no exposure to LARA, will use a standard wheelchair, and will be asked to perform a program of conventional arm exercises for 30 min/day, also in addition to standard of care rehabilitation therapy for 3 weeks or the duration of their stay.
  Other Names: Conventional Arm and Hand Exercise Program
  Arms: The Standard Therapy

SUMMARY:
This study will test the effectiveness of a new lever drive wheelchair, LARA - Lever Actuated Resonance Assistance. LARA facilitates patients in performing a high amount of practice using their moderate to severely impaired upper extremity after stroke.

Investigators will recruit 44 subjects with subacute strokes to participate in the study through the acute rehabilitation unit of the UC Irvine Douglas Hospital. Study participants will be randomized into 2 groups: LARA therapy group or standard therapy group. The LARA therapy group will use LARA to propel themselves to therapy appointments in the unit and to play video games with the affected upper extremity for 30 mins / day. The standard therapy group will use a standard wheelchair to propel themselves using their unaffected upper and lower extremities. They will be asked to perform a matched duration of standard arm exercises for 30 mins/ day. This program of standard arm exercises was developed by an OT at the Rehabilitation Institute of Chicago which consists of graded-difficulty table-supported exercises.

This study will have 3 assessment visits: baseline, 3 weeks after therapy or upon discharge from the acute rehabilitation unit if sooner, and a 3-month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of enrollment
2. Stroke onset 1-4 weeks prior to study enrollment
3. Arm motor FM score of < 30 (out of 66) at Baseline Visit
4. Absence of moderate to severe shoulder pain ( Score <3 on the 10 point visual analog pain scale)
5. Any deficit in vision, alertness, language, attention, or other cognitive functions that interfere with playing the LARA games

Exclusion Criteria:

1. Age >80 years at the time of enrollment
2. Severe tone in the affected upper extremities (Score ≥ 4 on the Modified Ashworth Spasticity Scale)
3. Severe language problem that would prevent participants from properly understanding instructions
4. Severe reduced level of consciousness
5. Severe aphasia (score of 3 on the NIH stroke scale (question 9))
6. Severe loss of sensation in stroke-affected upper extremities (Score < 1 on the Nottingham sensory assessment)
7. Currently pregnant
8. Difficulty in understanding or complying with the instructions given by the experimenter
9. Inability to perform the experimental task that will be studied

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cramer, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith BW, Lobo-Prat J, Zondervan DK, Lew C, Chan V, Chou C, Toledo S, Reinkensmeyer DJ, Shaw S, Cramer SC. Using a bimanual lever-driven wheelchair for arm movement practice early after stroke: A pilot, randomized, controlled, single-blind trial. Clin Rehabil. 2021 Nov;35(11):1577-1589. doi: 10.1177/02692155211014362. Epub 2021 May 24. PMID 34027703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from June 2017 to May 2018.
Pre-assignment Details: 23 study participants were screened and all 23 study participants were randomized.
Period: Overall Study
Arm/Group | The LARA Therapy | The Standard Therapy
Started | 12 | 11
Completed | 11 | 8
Not Completed | 1 | 3
Not completed — Relocation to out of the country | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Discharged to SNF, no transportation. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The LARA Therapy | The Standard Therapy | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We did not include the 4 study participants who dropped out the study to analysis: 1 from the LARA group and 3 from the Standard Therapy group,
  years
    number analyzed (Participants) | 11 | 8 | 19
    (all) | 52.1 (7.9) | 52.6 (9.5) | 52.32 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer (FM) Motor Assessment of the Upper Extremity
Description: We measure the change of the Fugl-Meyer Motor Assessment scores from the baseline evaluation to the 3-month follow up evaluation after the end of intervention. Fugl-Meyer is a 66-point scale measuring the movement pattern of the upper extremities. For the study, we analyze the total score only. The higher scores indicate a better outcome.
Time Frame: Baseline, Post-intervention evaluation at 3 weeks, and 3-month evaluation after the end of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The LARA Therapy | The Standard Therapy
Number analyzed (Participants) | 11 | 8
score on a scale
  Baseline Evaluation | 28.5 (11.6) | 27.4 (14.7)
  Change in Post therapy Evaluation | 14.2 (10.8) | 7.9 (3.8)
  Change in 3-month post-intervention | 18.8 (12.5) | 14.1 (7.4)

2. Secondary Outcome: Modified Ashworth Spasticity Scale
Description: We measure the spasticity of the upper extremity at baseline, post-intervention, and at the 3-month follow up evaluation. Spasticity is described as the resistance to passive movement. Participants are asked to relax and evaluators assess muscle resistance to passive movement at one joint at a time: Shoulder, Elbow, Wrist, and Fingers. The evaluator will then grade the resistance on a 6-point scale for each joint. Higher scores indicate more rigid movement or more muscle tone resistance. The minimum score is zero and the maximum score is 4. For this study, we combine all subscores from each joint to compute a total spasticity score.
Time Frame: Baseline, Post-intervention evaluation at 3 weeks, and 3-months after the end of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The LARA Therapy | The Standard Therapy
Number analyzed (Participants) | 11 | 8
score on a scale
  Baseline Evaluation | 0.64 (0.64) | 0.56 (0.61)
  Post-Intervention Evaluation | 0.47 (0.56) | 0.77 (0.80)
  3-month Follow Up | 0.61 (0.72) | 0.96 (1.37)

3. Secondary Outcome: Timed 10-meter Walk
Description: We measure the time one takes to complete a 10-meter walk at baseline evaluation, the post-intervention evaluation, and the 3-month follow up evaluation. Participants are instructed to walk at a distance of 10-meter over a level surface with 2 meters for acceleration and 2 meters for deceleration. Participants are instructed to walk at their comfortable or normal speed over the entire distance. Participants are timed once the first foot passes the acceleration path; the time is stopped once the first foot enters the deceleration path. The lower scores indicate a better outcome.
Time Frame: Baseline, Post-intervention evaluation at 3 weeks, and 3-months after the end of intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | The LARA Therapy | The Standard Therapy
Number analyzed (Participants) | 11 | 8
Seconds
  Baseline Evaluation | 18.8 (9.7) | 23.4 (9.1)
  Post-Intervention Evaluation | 15.2 (7.5) | 14.4 (5.0)
  3-month Follow Up | 11.8 (4.4) | 11.8 (3.7)

4. Secondary Outcome: Box and Blocks Test
Description: We measured the Box and Blocks Test scores at baseline evaluation, the post-intervention, and at the 3-month follow up evaluation. Participants are instructed to move as many blocks as possible, one at a time, from one compartment in a box to a second compartment over a divider for a period of 60 seconds; each block that is moved is counted, and multiple blocks moved at the same time are counted are counted as a single block. The higher scores indicate a better outcome.
Time Frame: Baseline, Post-intervention evaluation at 3 weeks, and 3-months after the end of intervention
Measure: Mean (Standard Deviation); unit: blocks
Arm/Group | The LARA Therapy | The Standard Therapy
Number analyzed (Participants) | 11 | 8
blocks
  Baseline Evaluation | 8.5 (10.8) | 11.9 (13.6)
  Post-Intervention Evaluation | 23.5 (19.2) | 22.1 (22.7)
  3-month Follow Up | 53.4 (31.8) | 45.8 (44.6)

ADVERSE EVENTS:
Time Frame: From intervention up to 3-month evaluation after the end of the intervention.
Arm/Group | The LARA Therapy | The Standard Therapy
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
Early termination of the study due to the budgetary issue leading to a smaller number of subjects recruited and fewer secondary outcome measures collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT02830893/Prot_SAP_000.pdf